CLINICAL TRIAL: NCT05772715
Title: The THumb Osteoarthritis Exercise TriAl (THETA); a Multicenter, Randomized Controlled Trial on Exercise Therapy with an Orthosis Compared to an Orthosis Alone in Patients with Thumb Base Osteoarthritis
Brief Title: The THumb Osteoarthritis Exercise TriAl
Acronym: THETA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Xpert Clinics (Unknown); Franciscus Gasthuis (Other); IJsselland ziekenhuis (Unknown); Reinier Haga Orthopedisch Centrum (Other); Elisabeth-TweeSteden Ziekenhuis (Other)
Responsible Party: Principal Investigator, Dr. Robbert Wouters, Dr. Robbert Wouters, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 852002001
Record Dates: First submitted 2022-12-23; First posted 2023-03-16 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Thumb Osteoarthritis
Keywords: exercise; orthosis
MeSH Terms: conditions — Motor Activity | interventions — Orthotic Devices; Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Orthosis group (Active Comparator)
  Interventions: Other: Orthosis
- Orthosis + exercise group (Experimental)
  Interventions: Other: orthosis + exercise therapy

INTERVENTIONS:
Other: orthosis + exercise therapy — The orthosis + exercise group receives the same orthosis and instructions as the orthosis group (see next section), supplemented by exercise therapy. This includes weekly 25-30-minute physical therapy sessions with a total of 12 sessions. Sessions include patient education on thumb positioning, functional training and home exercise instructions to improve CMC-1 stability during pinch in extension/abduction, as instability and degeneration occurs in flexion/adduction(17,19,28-31). The first phase (week 0 - week 6) comprises coordination exercises for the thumb intrinsics (except adductor pollicis), extensor pollicis brevis and first dorsal interosseous to support CMC-1 extension/abduction. The second phase (week 6 - month 3) comprises reduced orthosis usage and thenar muscle strengthening exercises(except adductor pollicis).
  Arms: Orthosis + exercise group
Other: Orthosis — The orthosis group receives a custom-made thermoplastic orthosis immobilizing the first carpometacarpal joint (CMC-1) in extension/abduction and the metacarpophalangeal joint in flexion. Orthosis usage is 24/7 in the first two weeks, thereafter only during activities with high load until three months. Two appointments take place: one for orthosis fabrication and one for a one-week checkup.
  Arms: Orthosis group

SUMMARY:
THIS TRIAL WAS PROSPECTIVELY REGISTERED ON FEBRUARY 27, 2020 IN THE DUTCH TRIAL REGISTRY (www.trialregister.nl), BUT THIS TRIAL REGISTRY WAS TERMINATED. THE DATA ON OUR TRIAL WERE TRANSFERED BY THE DUTCH TRIAL REGISTRY TO WHO'S CLINICAL TRIALS SEARCH PORTAL (REFERENCE NUMBER: NL-OMON54664). WE ALSO REGISTERED THE TRIAL HERE AT CLINICALTRIALS.GOV TO BE ABLE TO ADD MORE DETAILS ON OUR STUDY.

Summary:

OBJECTIVE(S)/RESEARCH QUESTION(S) Does an orthosis combined with exercise therapy results in less pain and less conversion to surgery than an orthosis alone in patients with first carpometacarpal osteoarthritis (CMC-1 OA), at three months and one year after the start of treatment? HYPOTHESIS The investigators hypothesize that the orthosis + exercise therapy group has less pain and conversion to surgery will be lower than the orthosis group.

STUDY DESIGN Randomized controlled multicenter trial STUDY POPULATION(S)/DATASETS Patients with first carpometacarpal osteoarthritis (CMC-1 OA) seeking treatment INTERVENTION Orthosis + exercise therapy USUAL CARE/COMPARISON Orthosis only OUTCOME MEASURES Primary outcomes: pain and conversion to surgery SAMPLE SIZE CALCULATION/DATA ANALYSIS Two groups of 80 participants; analysis based on repeated measures analysis (for pain) and Chi-square tests (for conversion to surgery). The investigators initially planned to perform a survival analysis (log-rank) and logistic regression for conversion to surgery but decided prior to data analysis on using chi-square tests to determine whether there is a between-group difference in the proportion of conversion to surgery. The investigators made this decision due to low inclusion rates, as chi-square tests require smaller sample sizes. The investigators will use a mixed-effect model analysis for pain.

COST-EFFECTIVENESS ANALYSIS (CEA)/ BUDGET IMPACT ANALYSIS (BIA) Economic evaluation will be done from societal & healthcare perspectives, according cost-effectiveness analysis (CEA) guidelines. Medical & non-medical costs and consequences (i.e. productivity loss) will be collected and taken into account. Both CEA and cost-utility analysis will be performed, using conversion to surgery and Quality-adjusted life years (QALYs), respectively TIME SCHEDULE Start preparation: December 2019, inclusion: October 2020- December 2022, final report: December 2023

ELIGIBILITY:
Inclusion criteria: All participants must meet the following criteria: 1) aged 18 or older; 2) Eaton stage 2-4 first carpometacarpal osteoarthritis (CMC-1 OA) based on radiographics and/or clinical examination; and 3) ability to visit the treatment center for treatment sessions.

Exclusion criteria: A potential participant that meets any of the following criteria will be excluded: 1) secondary first carpometacarpal osteoarthritis (CMC-1 OA) (e.g., due Bennett's fracture); 2) presence of comorbidity that interferes with treatment or outcome (e.g., carpal tunnel syndrome or De Quervain tenosynovitis); 3) surgery in medical history that interferes with treatment or outcome (e.g., trapeziectomy or tendon repair); 4) steroid injection in hand/wrist <6 weeks prior to admission; 5) previous treatment for CMC-1 OA in one of both hands, including orthosis, hand therapy or surgery; or 6) insufficient ability to understand written and spoken Dutch or English language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Pain - change | 3 months (primary), other Time points: baseline, 6 weeks, 6 months, 1 year.
  Michigan Hand Outcomes Questionnaire
Conversion to surgical treatment | 12 months
  Questionnaire: surgery yes/no

SECONDARY OUTCOMES:
Health-related quality of life | Time points: baseline, 6 weeks, 3 months, 6 months, 1 year.
  EuroQol-5-Dimension-5-levels
Hand Function | Time points: baseline, 6 weeks, 3 months, 6 months, 1 year.
  Michigan Hand Outcomes Questionnaire
Satisfaction with treatment results | Time points: 6 weeks, 3 months, 6 months, 1 year.
  Satisfaction with Treatment Result Questionnaire
Return to work | Time points: 6 weeks, 3 months, 6 months, 9 months, 1 year.
  Return to work
Grip & Pinch strength | Time points: baseline, 6 weeks, 3 months, 6 months, 1 year.
  Hand-held dynamometer and Pinch
Range of motion | Time points: baseline, 6 weeks, 3 months, 6 months, 1 year.
  Goniometry and Kapandji Score
Experience with healthcare delivery | Time points: 6 weeks, 3 months.
  Patient Reported Experience Measure
Complications | Time points: baseline, 6 weeks, 3 months, 6 months, 1 year.
  ICHOM Modified Clavien-Dindo Classification
Costs and productivity loss | Time points: 6 weeks, 3 months, 6 months, 9 months, 1 year.
  Productivity Cost Questionnaire, Medical Consumption Questionnaire
Treatment adherence | Time points: 6 wks, 3 months
  Therapy Adherence Assessment Tool
Treatment credibility and expectations | Time points: baseline, 6 weeks.
  Credibility/Expectancy Questionnare
Perceived attention/quality of the relationship | Time points: 6 weeks, 3 months.
  Consultation and Relational Empathy Measure
Depression | Time points: baseline,3 months.
  Patient Health Questionnaire-9
Anxiety | Time points: baseline, 3 months.
  General Anxiety Disorder-7
Illness perception | Time points: baseline, 3 months.
  Brief Illness Perception Questionnaire
Pain catastrophizing | Time points: baseline.
  Pain Catasctriphizing Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ruud W Selles, PhD, Principal Investigator — Erasmus Medical Center
Locations (5):
- Netherlands (5):
  - Xpert Clinics (multiple sites), Eindhoven, North Brabant
  - Elizabeth-TweeSteden Ziekenhuis, Tilburg, North Brabant
  - IJsselland ziekenhuis, Capelle aan den IJssel, South Holland
  - Franciscus Gasthuis, Rotterdam, South Holland
  - Reinier Haga Orthopedisch Centrum, Zoetermeer, South Holland

IPD SHARING:
Plan to Share IPD: Yes
We will manage the data following FAIR principles and store the data in DANS

REFERENCES:
- [Derived] Wouters RM, Esteban Lopez LM, Heemskerk SC, Bierma-Zeinstra SM, Kraan GA, Colaris J, Zuidam JM, Vermeulen GM, Selles RW; THETA Study Group Collaborators. Effectiveness of exercise therapy in patients with thumb carpometacarpal osteoarthritis: A multicenter, randomized controlled trial. Osteoarthritis Cartilage. 2025 Oct 23:S1063-4584(25)01187-2. doi: 10.1016/j.joca.2025.10.005. Online ahead of print. PMID 41138847